CLINICAL TRIAL: NCT00734877
Title: UARK 2013-13, Total Therapy 4B - Formerly 2008-01 - A Phase III Trial for Low Risk Myeloma Ages 65 and Under: A Trial Enrolling Subjects to Standard Total Therapy 3 (S-TT3)
Brief Title: UARK 2013-13, Total Therapy 4B - Formerly 2008-01 - A Phase III Trial for Low Risk Myeloma
Acronym: TT4B
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103668
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Bortezomib; Thalidomide; Dexamethasone; Cisplatin; Doxorubicin; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A (Active Comparator): The standard TT3 Regimen (S-TT3) will consist of 2 cycles of induction therapy with M-VTD-PACE and PBSC collection after the 1st cycle. MEL-based tandem transplant will be administered 6 weeks to 3 months apart, applying single dose MEL 200 mg/m2 with adjustments for age and renal function. Consolidation will consist of 2 cycles of dose-reduced VTD-PACE. Maintenance treatment will employ VRD for 3 years.
  Interventions: Drug: M-VTD-PACE
- ARM B (Experimental): The TT3-LITE Regimen (L-TT3) will employ only 1 cycle of induction therapy with MVTD- PACE
  Interventions: Drug: TT3-LITE Regimen (L-TT3)

INTERVENTIONS:
Drug: M-VTD-PACE — 2 cycles of induction therapy with M-VTD-PACE and PBSC collection after the 1st cycle. MEL-based tandem transplant will be administered 6 weeks to 3 months apart, applying single dose MEL 200 mg/m2 with adjustments for age and renal function. Consolidation will consist of 2 cycles of dose-reduced VTD-PACE. Maintenance treatment will employ VRD for 3 years.
  Other Names: Melphalan; Velcade; Thalidomide; Dexamethasone; Cisplatin; Adriamycin; Cyclophosphamide; Etoposide
  Arms: ARM A
Drug: TT3-LITE Regimen (L-TT3) — The TT3-LITE Regimen (L-TT3) will employ only 1 cycle of induction therapy with MVTD-PACE and, as in S-TT3, PBSC collection following recovery from this one and only induction treatment. MEL-based tandem transplant will be administered 6 weeks to 3 months apart, applying fractionated MEL200mg/m2 in 4 successive daily fractions of 50mg/m2 (MEL50 x 4) with addition of VTD with adjustments for age and renal function. Consolidation will consist of only 1 cycle of dose-reduced VTD-PACE. Maintenance treatment will employ VRD for 3 years.
  Other Names: Velcade (bortezomib); Melphalan; Dexamethasone; Thalidomide; Cisplatin; Adriamycin; Cyclophosphamide; Etoposide
  Arms: ARM B

SUMMARY:
Toward improving the therapeutic index of standard TT3 (S-TT3), the investigators will employ a randomized Phase III trial design to determine whether S-TT3 treatment-related toxicities can be reduced by 50% in TT3-Lite (L-TT3).

Note: Randomization has been discontinued and accrual is closed to the L-TT3 arm. This trial is currently enrolling as a single-arm trial for patients to receive S-TT3.

DETAILED DESCRIPTION:
The major treatment-related toxicities in TT3 pertained to the high-dose melphalan 200mg/m2 (MEL200)-based tandem transplant approach, consisting of mucosal and other toxicities.

For the TT4 trial, we are proposing to compare standard TT3 (S-TT3) to TT3-Lite (L-TT3). L-TT3 will employ various strategies aimed at improving the therapeutic Index of S-TT3 by reducing toxicities while maintaining the superior results reported for S-TT3 in terms of frequency and duration of CR, EFS, and. The following strategies will be utilized in L-TT3:

* Applying only 1 instead of 2 cycles of induction and consolidation therapy prior to and after tandem transplant. This is supported by the well known association between prior exposure to mucotoxic therapies4, 5 and worse post-transplant mucositis, particularly when etoposide is used in the mobilizing regimen6 such as in VDTPACE.

Note: Randomization has been discontinued and accrual is closed to the L-TT3 arm. This trial is currently enrolling as a single-arm trial for patients to receive S-TT3.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed active MM requiring treatment. Patients with a previous history of smoldering myeloma will be eligible if there is evidence of progressive disease requiring chemotherapy.
* Patients must be either untreated or have not had more than one cycle of systemic MM therapy, excluding bisphosphonates and localized radiation.
* Participants must have low-risk disease, as defined by any of the following:

  * GEP risk score of < 0.66
  * lack of GEP-defined TP53 deletion (Affymetrix signal <727)
  * No metaphase based abnormalities of 1q or 1p
  * LDH <360 U/L Rule out hemolysis, infection, and contact PI for Clarification
* Zubrod ≤ 2, unless solely due to symptoms of MM-related bone disease.
* Patients must be at least 18 years of age and not older than 75 years of age at the time of registration.
* Participants must have preserved renal function as defined by a serum creatinine level of < 3 mg/dL.
* Participants must have an ejection fraction by ECHO or MUGA ≥ 40%
* Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) > 50% of predicted. If the patient is unable to complete pulmonary function tests due to MM related pain or condition, exception may be granted if the principal investigator documents that the patient is a candidate for high dose therapy.
* Patients must have signed an IRB-approved informed consent indicating their understanding of the proposed treatment and understanding that the protocol has been approved by the IRB.

Exclusion Criteria:

* High risk disease defined by high-risk gene array features as determined by any of the following:

  * GEP risk score of ≥ 0.66 or
  * Presence of GEP-defined TP53 deletion, or
  * Presence of abnormalities of chromosome 1 (amp1q, del 1p).
* Poorly controlled hypertension, diabetes mellitus, or other serious medical illness or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Platelet count < 30 x 109/L, unless myeloma-related.
* Grade > 2 peripheral neuropathy.
* Hypersensitivity to bortezomib, boron, or mannitol.
* Recent (< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias.
* Evidence of chronic obstructive or chronic restrictive pulmonary disease.
* Patients must not have light chain deposition disease or creatinine > 3 mg/dl
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for at least three years. Prior malignancy is acceptable provided there has been no evidence of disease within the three-year interval or if the malignancy is considered much less life threatening than the myeloma.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | 3 years from study enrollment
  Percentage of subjects without disease progression (per IMWG definition) at 3 years from initial registration

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Zangari, MD, Principal Investigator — UAMS; Maurizio Zangari, MD, Study Director — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Myeloma Institute for Research and Therapy, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Ling W, Zangari M, Van Rhee F, Barlogie B, Yaccoby S. Altered mesenchymal and endothelial subsets in interstitial bone marrow and focal lesions in myeloma patients and SCID-hu mice. Haematologica. 2025 Nov 1;110(11):2740-2751. doi: 10.3324/haematol.2025.287717. Epub 2025 Jun 12. PMID 40501401
- [Derived] Davies FE, Rosenthal A, Rasche L, Petty NM, McDonald JE, Ntambi JA, Steward DM, Panozzo SB, van Rhee F, Zangari M, Schinke CD, Thanendrarajan S, Walker B, Weinhold N, Barlogie B, Hoering A, Morgan GJ. Treatment to suppression of focal lesions on positron emission tomography-computed tomography is a therapeutic goal in newly diagnosed multiple myeloma. Haematologica. 2018 Jun;103(6):1047-1053. doi: 10.3324/haematol.2017.177139. Epub 2018 Mar 22. PMID 29567784
- [Derived] Usmani SZ, Heuck C, Mitchell A, Szymonifka J, Nair B, Hoering A, Alsayed Y, Waheed S, Haider S, Restrepo A, Van Rhee F, Crowley J, Barlogie B. Extramedullary disease portends poor prognosis in multiple myeloma and is over-represented in high-risk disease even in the era of novel agents. Haematologica. 2012 Nov;97(11):1761-7. doi: 10.3324/haematol.2012.065698. Epub 2012 Jun 11. PMID 22689675
- See also: UAMS Myeloma Center — https://cancer.uams.edu/myeloma/